CLINICAL TRIAL: NCT06649604
Title: Alleviating Panretinal Photocoagulation Associated Ocular Pain With Vibratory Stimulation
Brief Title: Reducing Pain From Retinal Laser With Vibrational Stimulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Retina Consultant (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00144813
Record Dates: First submitted 2024-10-07; First posted 2024-10-21 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Pain, Perioperative
Keywords: Vibration Anesthesia Device; Perioperative Pain Alleviation; Panretinal Photocoagulation; Diabetic retinopathy treatment
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: All patient are their own control, using laser in both eyes, but only one using the Vibration Anesthesia Device.
Who Masked: Outcomes Assessor
Masking Description: Only the collaborator who will analyse the data will be masked, due to the manifest presence or absence of the vibratory device for both the clinician and the patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PRP with the Vibration Anesthesia Device (Experimental): Laser for PRP treatment as usual, but with the addition of the Vibration Device in one of the two eyes of a patient (The other eye receiving the same laser treatment without the device).
  Interventions: Device: Vibration Anesthesia Device; Procedure: Panretinal Photocoagulation
- PRP without the Vibration Anesthesia Device (Active Comparator): Laser for PRP treatment as usual in one of the two eyes of a patient (other eye receiving the same treatment, but with the Vibration Device).
  Interventions: Procedure: Panretinal Photocoagulation

INTERVENTIONS:
Device: Vibration Anesthesia Device — The intervention arm of this study is distinguished by way of the use of the Vibration Anesthesia Device
  Arms: PRP with the Vibration Anesthesia Device
Procedure: Panretinal Photocoagulation — Laser treatment for diabetic retinopathy done in a standard fashion

SUMMARY:
The goal of this clinical trial is to learn if Vibration Anesthesia Device works to reduce pain during retinal laser for diabetic retinopathy. The main question it aims to answer is:

Does the Vibration Anesthesia Device reduces the pain felt by patients during the laser treatment? Researchers will compare the standard method (no vibration device) to the standard method with the Vibration Anesthesia Device to see if the device works to reduce discomfort during treatment.

Eligible participants will have both eyes treated as required, one eye with the device and the other one without. Both the side that will be treated with the device in place and the first side to be treated will be decided by random sequence.

DETAILED DESCRIPTION:
Background:

Panretinal photocoagulation (PRP) is a widely used laser treatment for proliferative diabetic retinopathy (PDR). However, the associated ocular pain can make the procedure uncomfortable, leading to increased treatment visits or missed appointments. This pain is multifactorial and can be exacerbated by factors such as anxiety and hypervigilance. Traditional pain management techniques, such as regional anesthesia, are effective but invasive and carry potential complications. Oral medications have largely proven ineffective in alleviating PRP-related pain.

The Gate-Control Theory of pain posits that non-noxious stimuli can inhibit pain signals by activating A-β fibers, effectively "closing the gate" to pain transmission through A-δ and C fibers. The most relatable example is the mother rubbing a child's knee after an impact injury in the affected region. Transcutaneous electrical nerve stimulation (TENS) which utilizes the Gate-Control Theory of pain, has been shown to reduce ocular pain during PRP. However, its use raises practical concerns, including the need to carefully adjust pulse width, intensity, and frequency for effective pain relief. Additionally, some patients may find the muscular contractions or paresthesia uncomfortable. TENS is also contraindicated in individuals who are pregnant, have epilepsy, or have pacemakers. Vibratory stimulation activates cutaneous mechanoreceptors to reduce pain during intramuscular and subcutaneous injections. This technique is safer and less invasive than TENS and is therefore an ideal candidate for evaluating its effect in pain reduction during PRP. This study has the potential for an innovative concept by utilizing a vibratory device integrated within the PRP machine headrest.

Hypothesis:

Vibratory stimulation is expected to reduce ocular pain during PRP by activating cutaneous mechanoreceptors and inhibiting pain transmission, as suggested by the Gate-Control Theory. Its non-invasive nature makes it a practical alternative to traditional pain management methods, potentially enhancing patient comfort during the procedure.

Objective:

To evaluate the effectiveness of vibratory stimulation in reducing ocular pain during PRP treatments

Method:

Subjects will be recruited at a single tertiary referral center (Alberta Retina Consultants, Edmonton, Alberta). Matriculation will be established upon obtainment of consent, and patients will have the autonomy to withdraw from the study at any stage. The enrollment period will be from October 2024 to March 2025, with a total of 50 patients.

Laser settings will be tailored to each patient based on individual differences in pigmentation and tissue uptake. The threshold for treatment will be determined by observing an opacified photothermic response. For each patient, one eye will be treated without vibratory stimulation, while the contralateral eye will receive stimulation using the Blaine Labs Vibration Anesthesia Device. The assignment of which eye receives which treatment will be randomized using Python programming, ensuring a balanced allocation. To minimize variability, the time taken to perform PRP on both eyes will be kept as equal as possible. A no-treatment zone of 1 clock hour from the horizontal meridian will be maintained to avoid the long ciliary nerves. After treatment, patients will complete a validated survey based on the numeric rating scale (NRS) to assess pain levels for each eye treated.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve patients
* Bilateral PRP for proliferative diabetic retinopathy required
* >500 applications to each eye
* < 51 applications difference between each eye, in the superior or inferior hemisphere.

Exclusion Criteria:

* Poor pupil dilation < 5mm
* Media opacity preventing laser

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-10-15 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Pain Rating Scale | At time of enrolment
  Patient are enrolled on the same day as the study treatment. Patients will rate their pain sensation. They will have their first eye (left or right and with or without the Anesthesia Vibration Device based on randomization) treated, then they will assess their pain sensation. After this assessment, during the same session, their second eye will be treated and they will be asked to complete the same assessment for this second eye. The provided form to assess this outcome is a numeric scale from 0 (no pain) to 10 (worst possible pain) using the Wong-Baker Faces scale.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Tennant, MD, FRCSC, Principal Investigator — University of Alberta
Locations (1):
- Alberta Retina Consultant, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No